CLINICAL TRIAL: NCT03924544
Title: Decorin as an Antifibrotic Agent in Sub Scleral Trabeculectomy: A Pilot Study
Brief Title: Decorin in Sub Scleral Trabeculectomy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Collaborators: University of Luebeck (Other)
Responsible Party: Principal Investigator, abdussalam abdullatif, MD, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0321
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Primary Open-angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Decorin; Mitomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decorin Group (Experimental): 26 patients will receive subconjunctival injection of 100 µg decorin 15 minutes before surgery, 1, 3, and 7postoperatively. A30-gauge needle was used to inject 100 µL of decorin. The needle was placed at the nasal margin of the superior rectus muscle
  Interventions: Drug: Decorin
- Mitomycin Group (Active Comparator): MMC will then be applied in 26 patients to the sclera at a concentration of 0.3 mg/ml using cellulose sponges, which will be removed after 3 minutes followed by copious irrigation with balanced saline solution (BSS).
  Interventions: Drug: Mitomycin c

INTERVENTIONS:
Drug: Decorin — Antifibrotic agent
  Arms: Decorin Group
Drug: Mitomycin c — Antifibrotic agent
  Arms: Mitomycin Group

SUMMARY:
This is a prospective, single-center, interventional, randomized controlled study comparing Decorin as antifibrotic agent in sub scleral trabeculectomy versus Mitomycin.

DETAILED DESCRIPTION:
Study design:

This is a prospective, single-center, interventional, randomized controlled study at Kasr Al Aini Teaching Hospital, Cairo University. Patients with medically uncontrolled glaucoma will be enrolled in our study.

Fifty two consecutive eyes with Primary Open-angle Glaucoma indicated for trabeculectomy will be enrolled in the current study and will be then randomly assigned to our interventions. Informed consent will be obtained from all patients before any intervention. Uncontrolled glaucoma was defined as uncontrolled IOP (≥22 mm Hg) measured with a Goldmann applanation tonometer under maximal tolerable medical treatment with visual field defect progression. Exclusion criteria will include patients with history of intraocular surgery within the previous 6 months, patients with history of surgery involving the conjunctiva, angle closure glaucoma, and patient refusal to take part in the study.

Data Collected:

Preoperative:

Preoperative information that will be collected will include the patient's age, sex, previous ocular procedures, number of glaucoma medications, last recorded intraocular pressure (IOP), ocular comorbidity, and best corrected visual acuity (VA).

Adjuvant Decorin:

Recombinant human decorin will be provided by the manufacturing company (R&D Systems, Inc., Minneapolis, MN, USA) reconstituted in a vial at 0.4% concentration using phosphate-buffered saline as a vehicle.

Surgical Procedure:

In Decorin group: 26 patients will receive subconjunctival injection of 100 µg decorin 15 minutes before surgery. A30-gauge needle was used to inject 100 µL of decorin. The needle was placed at the nasal margin of the superior rectus muscle, so that a visible bleb was formed on the supranasal quadrant.

A corneal traction suture will be taken, followed by fornix-based conjunctival dissection and gentle diathermy.

Mitomycin Group: MMC will then be applied in 26 patients to the sclera at a concentration of 0.3 mg/ml using cellulose sponges, which will be removed after 3 minutes followed by copious irrigation with balanced saline solution (BSS).

A half to three-quarter thickness, rectangular scleral flap will be dissected. Four grooves will be created into clear cornea near the limbus to accommodate the releasable sutures then two preplaced releasable sutures will be taken at the corners of the scleral flap using 10/0 nylon sutures. The corneal traction will then be released and the trabeculectomy ostium will be created using a 0.75 mm Kelly's punch (Katena Products Inc., Denville, NJ) followed by a peripheral iridectomy (PI). The two releasable sutures will be tied, and BSS was used to form the anterior chamber. More releasable sutures will be taken in the middle of the scleral flap until watertight closure is achieved. The conjunctival incision will then be closed by 2 purse string sutures at the sides and one mattress suture at the limbus, using 10/0 nylon sutures.

Topical prednisolone 1% eyedrops will be used every 2 hours for 2 weeks, 6 times daily for 2 weeks, then tapered gradually over the following 2 months. Topical moxifloxacin 0.5% will be given 5 times daily for 2 weeks.

In Decorin group: postoperative days 1, 3, and 7, patients will receive subconjunctival injection of decorin. A30-gauge needle was used to inject 100 µL of decorin at the nasal margin of the superior rectus muscle.

Postoperative:

Patients will be seen after 1 day, 1 week, 1 month, 3 months, 6 months, 9 months and 12 months, with more frequent visits in uncontrolled or complicated cases. IOP and visual acuity measurements will be recorded every visit. Any complications of surgery will be reported.

Primary outcome measure is success of trabeculectomy defined as complete if the IOPis≤ 21 mm Hg without medications and qualified where antiglaucoma therapy is required to maintain it at such a level. Failure will be defined as an IOP> 21 mmHg on medications, need for another glaucoma surgery or loss of light perception.

.

ELIGIBILITY:
Inclusion Criteria:

* Primary Open Angle Glaucoma

Exclusion Criteria:

* Secondary Glaucoma, Closed angle glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
success of trabeculectomy | one year
  complete if the IOPis≤ 21 mm Hg without medications

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdullatif AM, Macky TA, Abdullatif MM, Nassar K, Grisanti S, Mortada HA, Soliman MM. Intravitreal decorin preventing proliferative vitreoretinopathy in perforating injuries: a pilot study. Graefes Arch Clin Exp Ophthalmol. 2018 Dec;256(12):2473-2481. doi: 10.1007/s00417-018-4105-7. Epub 2018 Aug 20. PMID 30128605
- [Background] Grisanti S, Szurman P, Warga M, Kaczmarek R, Ziemssen F, Tatar O, Bartz-Schmidt KU. Decorin modulates wound healing in experimental glaucoma filtration surgery: a pilot study. Invest Ophthalmol Vis Sci. 2005 Jan;46(1):191-6. doi: 10.1167/iovs.04-0902. PMID 15623773
- [Background] Nassar K, Luke J, Luke M, Kamal M, Abd El-Nabi E, Soliman M, Rohrbach M, Grisanti S. The novel use of decorin in prevention of the development of proliferative vitreoretinopathy (PVR). Graefes Arch Clin Exp Ophthalmol. 2011 Nov;249(11):1649-60. doi: 10.1007/s00417-011-1730-9. Epub 2011 Jul 7. PMID 21735240